CLINICAL TRIAL: NCT01482195
Title: Phase I Trial of Ocular Subretinal Injection of a Recombinant Adeno-Associated Virus (rAAV2-VMD2-hMERTK) Gene Vector to Patients With Retinal Disease Due to MERTK Mutations
Brief Title: Trial of Subretinal Injection of (rAAV2-VMD2-hMERTK)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: King Khaled Eye Specialist Hospital (Other Government)
Collaborators: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0916-P
Record Dates: First submitted 2011-09-28; First posted 2011-11-30 (Estimated); Results first posted 2021-07-15 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Retinal Disease; Retinitis Pigmentosa
Keywords: Retinal Disease; subretinal gene therapy; MERTK; retinitis pigmentosa
MeSH Terms: conditions — Retinal Diseases; Retinitis Pigmentosa

STUDY DESIGN:
Intervention Model Description: Ocular Subretinal administration of rAAV2-VMD2-hMERTK .
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subretinal Injection of rAAV2-VMD2-hMERTKRecombinant Adeno-Associated Virus (Experimental): Single arm of 6 patients undergoing subretinal injection of Gene Therapy using rAAV2-VMD2-hMERTKRecombinant Adeno-Associated Virus. Each patient received the injection in one eye.
  Interventions: Biological: Subretinal administration of rAAV2-VMD2-hMERTKRecombinant Adeno-Associated Virus
- fellow eye without intervention (No Intervention): fellow eye without intervention

INTERVENTIONS:
Biological: Subretinal administration of rAAV2-VMD2-hMERTKRecombinant Adeno-Associated Virus — The study is an open-label, dose-escalation, phase I clinical trial of subretinal administration of rAAV2-VMD2-hMERTK in patients with retinitis pigmentosa due to MERTK mutation.
  Arms: Subretinal Injection of rAAV2-VMD2-hMERTKRecombinant Adeno-Associated Virus

SUMMARY:
This study was to assess the safety of gene transfer via subretinal administration of rAAV2-VMD2-hMERTK in subjects with MERTK-associated retinitis pigmentosa (RP).

DETAILED DESCRIPTION:
In this phase I open-label, dose-escalation trial, one eye of each patient (the worse-seeing eye in five subjects) will receive a submacular injection of the subretinal rAAV2-VMD2-hMERTK. Patients will be followed daily for 10 days and then at 30, 60, 90, 180, 270, 365, 540, and 730 days post-injection. Data will be collected on (1) full ophthalmologic examination including best-corrected VA, intraocular pressure, color fundus photographs, macular spectral-domain optical coherence tomography, and full-field stimulus threshold test (FST) in both the study and fellow eyes; (2) systemic safety data including CBC, liver, and kidney function tests, coagulation profiles, urine analysis, AAV antibody titers, peripheral blood PCR and ASR measurement; and (3) listing of ophthalmological or systemic adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* MERTK-associated retinal disease;
* VA: 20/100 or less in worse eye
* Ability to perform tests of visual and retinal function;
* Good general health based on a complete physical examination and hematology and chemistry studies performed at a pre-treatment evaluation;
* Ability to comply with research procedures;

Exclusion Criteria:

* Pre-existing eye conditions that would preclude the planned surgery or interfere with the interpretation of study endpoints or surgical complications (for example, glaucoma, corneal or lenticular opacities);
* Complicating systemic diseases (such as medical conditions causing immunosuppression) that would preclude the gene transfer, ocular surgery or known sensitivity or allergy to medications planned for use in the peri-operative period;
* Use of anti-platelet agents that may alter coagulation within 7 days prior to study agent administration;
* Use of immunosuppressive medications;
* Pregnancy or breastfeeding;
* Individuals (males and females) of childbearing potential who are unwilling to use effective contraception for 1 year following agent administration and barrier contraception for 3 months following agent administration;
* Any other condition that would prevent a subject from completing follow-up examinations during the course of the study and that, in the opinion of the investigator, makes the subject unsuitable for the study.
* Current, or recent (within the past 30 days, or 10 half lives of the drug) participation, in any other research protocol involving investigational agents or therapies.
* Recent (within past 6 months) receipt of an investigational biologic therapeutic agent.Subjects will not be excluded based on their gender, race or ethnicity.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fowzan S Alkuraya, MD, Principal Investigator — King Faisal Specialist Hospital & Research Center
Locations (1):
- King Khaled Eye Specialist Hospital, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Wang CY, Chen L, Lin TY, Huang SP. Systematic Identification of Candidate Genes for Inherited Retinal Disease Gene Therapy Integrating Worldwide IRD Cohort and Single-Cell Analysis. J Ophthalmol. 2025 Jun 12;2025:7014745. doi: 10.1155/joph/7014745. eCollection 2025. PMID 40547876
- [Derived] Parinot C, Nandrot EF. A Comprehensive Review of Mutations in the MERTK Proto-Oncogene. Adv Exp Med Biol. 2016;854:259-65. doi: 10.1007/978-3-319-17121-0_35. PMID 26427420

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Six eyes of 6 patients were enrolled in this phase of the study. All patients had the typical clinical signs and symptoms of retinitis pigmentosa and tested positive for MERTK mutation. All patients were recruited from the outpatient clinics at King Khaled Eye specialist Hospital (KKESH) starting September 2011.
Groups:
- Recombinant Adeno-Associated Virus: Recombinant Adeno-Associated Virus: Ocular Subretinal Injection of a Recombinant Adeno-Associated Virus
Period: Overall Study
Arm/Group | Recombinant Adeno-Associated Virus
Started | 6
One Year Results | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Recombinant Adeno-Associated Virus
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 33.3 [14 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Region of Enrollment [Number; unit: participants]
  Saudi Arabia | 5
  Bahrain | 1

OUTCOME MEASURES:

1. Primary Outcome: Systemic and Ocular Safety
Description: Detailed history & physical exam were obtained at baseline visit and each post-injection protocol visit searching for systemic adverse events. Included were electrocardiogram, chest X-ray, complete blood count & differential, prothrombin time & INR, partial thromboplastin time, serum electrolytes, full serum chemistries including liver and renal function, urinalysis; serum antibody titers to AAV2 capsid components and antigen-specific reactivity (ASR) assays; blood analysis by DNA PCR to detect vector spread.
  Ophthalmic safety monitored changes from baseline included 1) corneal abnormalities, afferent pupillary defect, intraocular inflammation, cataract & intraocular pressure changes; 2) retinal changes based on fundus photos; 3) Macular SD-OCT changes in Central macular (CMT) and central foveal thickness (CFT) measurements when patient fixation allowed it, and 4) full field stimulus threshold (FST) to detect any retinal toxicity .
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Recombinant Adeno-Associated Virus Injected Eyes: Eyes with RP which received a single dose of subretinal recombinant Adeno-Associated Virus injection.
- Fellow Eyes: Eyes with RP which did not receive subretinal recombinant Adeno-Associated Virus injection.
Arm/Group | Recombinant Adeno-Associated Virus Injected Eyes | Fellow Eyes
Number analyzed (Participants) | 6 | 6
Participants
  Systemic events | 0 | 0
  Corneal abnormalities | 1 | 0
  Afferent pupillary defect | 0 | 0
  Intraocular inflammation | 0 | 0
  Cataract | 1 | 0
  Intraocular pressure changes | 0 | 0
  Retinal changes | 2 | 2
  Macular thinning on OCT | 0 | 1
  Toxicity seen on FST | 0 | 0

2. Secondary Outcome: Visual Acuity Measurement
Description: Although candidates may have very severe loss of function, an attempt was made to measure a best-corrected visual acuity using Early Treatment Diabetic Retinopathy Study (ETDRS) charts, and measurements were recorded as the number of letters read on each line of the chart (Diabetic Retinopathy Study Research Group 1985). If a patient was unable to read at least three letters of the first line correctly, the chart distance was progressively halved from the standard 4 m until either the first line was correctly read or the shortest distance of 0.5 m was reached. Patients who were unable to read any letters on the chart were tested for light perception and if they perceived light they were assigned the acuity score equivalent of <20/6400. Measurements were performed at baseline and each protocol follow up visit. Improvement in patients who could read was defined as a gain in 5 letters, and in those with those LP vision only to start seeing hand motion.
Time Frame: 2 years and up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Adeno-Associated Virus Injected Eyes | Fellow Eyes
Number analyzed (Participants) | 6 | 6
Participants
  Improved VA at 2 years | 3 | 1
  Decreased VA at 2 years | 0 | 2
  Stable VA at 2 years | 3 | 3
  Improvement of VA after 2years | 0 | 0

3. Secondary Outcome: Full-field Stimulus Threshold Testing (FST).
Description: Full-field stimulus threshold testing (FST) measures sensitivity of the entire visual field by estimating the lowest luminance of a flash that elicits a visual sensation. The FST measurements were performed at baseline and throughout the protocol visits over two years in the study and fellow eyes, and changes in FST results were analyzed.
Time Frame: 2 years
Population: Six Patients with the clinical diagnosis of RP with a proven MERTK mutation were included. Patients had to be older than 14 years of age and had the viral vector injected into their worse seeing one eye (except case #4).
Measure: Mean (95% Confidence Interval); unit: dB
Arm/Group | Recombinant Adeno-Associated Virus Injected Eyes | Fellow Eyes
Number analyzed (Participants) | 6 | 6
dB
  FST at baseline | -23.34 [-29.65 to -17.03] | -24.14 [-30.40 to -17.88]
  FST at 10 days | -19.58 [-25.93 to -13.23] | -20.13 [-26.59 to -13.67]
  FST at 30 days | -19.22 [-23.98 to -14.46] | -23.40 [-30.60 to -16.29]
  FST at 90 days: number analyzed (Participants) | 5 | 6
  FST at 90 days | -13.94 [-42.96 to 15.08] | -24.68 [-33.54 to -15.82]
  FST at 180 days: number analyzed (Participants) | 4 | 6
  FST at 180 days | -20.01 [-28.12 to -11.90] | -22.02 [-31.83 to -12.21]
  FST at 365 days: number analyzed (Participants) | 5 | 6
  FST at 365 days | -20.59 [-30.09 to -11.08] | -22.26 [-28.87 to -15.65]
  FST at 1.5 year: number analyzed (Participants) | 5 | 6
  FST at 1.5 year | -21.09 [-29.04 to -13.14] | -21.66 [-29.81 to -13.51]
  FST at 2 years: number analyzed (Participants) | 3 | 6
  FST at 2 years | -20.38 [-28.54 to -12.23] | -15.92 [-29.78 to -2.05]

4. Secondary Outcome: Central Foveal Thickness (CFT) on Optical Coherence Tomography (OCT).
Description: Central foveal thickness (CFT) measurements were performed at baseline and throughout the protocol visits over two years in the study and fellow eyes (whenever possible), and changes in CFT values were analyzed.
Time Frame: 2 years
Measure: Mean (95% Confidence Interval); unit: microns.
Arm/Group | Recombinant Adeno-Associated Virus Injected Eyes | Fellow Eyes
Number analyzed (Participants) | 5 | 5
microns.
  CFT at Baseline | 65.80 [36.69 to 94.91] | 74.80 [41.22 to 108.38]
  CFT at 2 years | 69.20 [39.89 to 98.51] | 75.00 [50.51 to 99.49]

5. Secondary Outcome: Central Macular Thickness (CMT) on Optical Coherence Tomography (OCT).
Description: Central macular thickness (CMT) measurements were performed at baseline and throughout the protocol visits over two years in the study and fellow eyes (whenever possible), and changes in CMT values were analyzed.
Time Frame: 2 years
Measure: Mean (95% Confidence Interval); unit: microns.
Arm/Group | Recombinant Adeno-Associated Virus Injected Eyes | Fellow Eyes
Number analyzed (Participants) | 3 | 3
microns.
  CMT at baseline | 128.00 [65.75 to 190.25] | 132.67 [40.56 to 224.76]
  CMT at 2 years | 132.33 [70.76 to 193.90] | 123.76 [48.92 to 198.41]

ADVERSE EVENTS:
Time Frame: through study completion, an average of 2 years
Description: The adverse events were collected :
  1. systematically ( blood samples withdrawn to test for rise in antiViral titers). One temporary rise occurred in the post-operative period in one patient = non serious adverse events)
  2. Non systematic collection: ( one patient reported filamentary keratitis, another patient eported oscillopsiain the injected eye- = Other non serious adverse events
Arm/Group | Recombinant Adeno-Associated Virus
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Adeno-Associated Virus (N=6)
Filamentary keratitis (Eye disorders) | 1 (1) — resolved with postoperative lubrication therapy
delayed resolution of subretinal fluid postoperatively, cataract, oscillopsia (Eye disorders) | 1 (1) — The fluid resolved spontaneously within 6 weeks after surgery with return of vision to baseline. The same patient developed posterior subcapsular cataract and persistent oscillopsia in the operated eye and the cause remains unknown.
systemic (Blood and lymphatic system disorders) | 1 (1) — One patient developed a rise in AAV antibodies but with a negative PCR. Serum AAV antibody and antigen specific reactivity measurements for the remaining patients are negative

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No